CLINICAL TRIAL: NCT02845713
Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Single Dose Treatment With Diethylcarbamazine, Albendazole and Ivermectin in Humans With and Without Wuchereria Bancrofti Infection in Côte d'Ivoire
Brief Title: Pharmacokinetics & Pharmacodynamics of Diethylcarbamazine (DEC)+ Albendazole (ALB) + Ivermectin (IVE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Christopher L. King, MD, PhD, Professor of International Health, Medicine and Pathology, Case Western Reserve University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 03-16-09
Record Dates: First submitted 2016-06-03; First posted 2016-07-27 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Wuchereria Bancrofti Infection
MeSH Terms: conditions — Elephantiasis, Filarial | interventions — Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single IDA dose W. bancrofti positive (Active Comparator): Single oral dose of Ivermectin, Diethylcarbamazine Albendazole (IDA) W. bancrofti infections positive
  Interventions: Drug: Ivermectin, Diethylcarbamazine Albendazole (IDA)
- Single IDA dose W. bancrofti negative (Active Comparator): Single oral dose of Ivermectin, Diethylcarbamazine Albendazole (IDA) in 40 individuals who are free of W. bancrofti infection.
  Interventions: Drug: Ivermectin, Diethylcarbamazine Albendazole (IDA)

INTERVENTIONS:
Drug: Ivermectin, Diethylcarbamazine Albendazole (IDA) — To evaluate the safety and tolerability of triple drug therapy (a single dose of ALB, IVM and DEC)
  Other Names: IDA

SUMMARY:
The study will be an open label cohort study with 2 two-treatment groups 2). Both groups will be treated with a single oral administration of Diethylcarbamazine (DEC) 6 mg/kg + Albendazole (ALB) 400 mg + Ivermectin (IVR) 200 µg/kg (IDA). One treatment group will include men and women with W. bancrofti infections (>50 Mf/ml, N=30). The other treatment group will include men and women who are free of W. bancrofti infection based on negative blood tests for both microfilariae (Mf) and circulating filarial antigen (N=30). Active follow-up for adverse events (AE) will be for 72hrs and passive follow-up for 7 days following treatment.

Participants will be followed again at 1 year to evaluate treatment efficacy. Individuals with severe AEs (grade 3 or higher) will be transported to the Agboville District Hospital and cared for by the hospital staff. Based on treatment of over 100 Lymphatic filariasis (LF) infected individuals any AEs develop within the first 72 hours following treatment and uncommonly up to 7 days post-treatment.

All individuals will be admitted to a single health center or hospital in Côte d'Ivoire.

Subjects will be monitored for 72-hours after treatment for safety and to facilitate sampling for drug analyses and safety tests. Participants will undergo clinical monitoring every 6 hours to evaluate potential adverse effects of Ivermectin + Diethylcarbamazine + Albendazole (IDA) treatment. Participants will also be monitored for hematologic, or biochemical abnormalities during the period of observation.

DETAILED DESCRIPTION:
The study will be an open label cohort study with 2 two-treatment groups. Both groups will be treated with a single oral administration of DEC 6 mg/kg + ALB 400 mg + IVR 200 µg/kg (IDA). One treatment group will include men and women with W. bancrofti infections (>50 Mf/ml, N=30). The other treatment group will include men and women who are free of W. bancrofti infection based on negative blood tests for both microfilariae and circulating filarial antigen (N=30). Active follow-up for adverse events (AE) will be for 72 hours and passive follow-up for 7 days following treatment.

Participants will be followed again at 1 year to evaluate treatment efficacy. Individuals with severe AEs (grade 3 or higher) will be transported to the Agboville District Hospital and cared for by the hospital staff. Based on treatment of over 100 LF infected individuals any AEs develop within the first 72 hours following treatment and uncommonly up to 7 days post-treatment.

All individuals will be admitted to a single health center or hospital in Côte d'Ivoire.

Subjects will be monitored for 72-hours after treatment for safety and to facilitate sampling for drug analyses and safety tests. Participants will undergo clinical monitoring every 6 hours to evaluate potential adverse effects of IDA treatment. Participants will also be monitored for hematologic, or biochemical abnormalities during the period of observation.

At enrollment all subjects will be otherwise healthy adult men and women (≥18-65 years of age). All individuals will be assessed for the presence and burden of geohelminth infections, parasitic worms of the gastrointestinal tract such as hookworm, Trichuris trichiuria and Ascaris lumbricoides. This is important because two of the drugs in the combination (ALB and IVM) are active against geohelminths. Individuals with heavy geohelminth burdens may experience adverse reactions because of rapid killing of their intestinal parasites.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide informed consent to participation in the study

  * Male or female 18-65 years of age
  * Peripheral blood microfilaremia levels >50 microfilaria/ml (treatment group 1)
  * No evidence of filarial infection by Mf and Circulating filarial antigen (CFA) testing (treatment group 2)
  * No history of taking anti-filarial medications in past 2 years

Exclusion Criteria:

Known chronic illness, e.g. tuberculosis, diabetes, renal insufficiency

* Anemia (Hb <7 g/dl) by HemaCue
* Not willing or able to give informed consent for the study
* Onchocerciasis rapid test (Ov16) and/or skin snip positive for onchocerciasis
* Permanent disability that prevents or impedes study participation and/or comprehension Pregnancy. Women will be tested with a rapid urine test for beta human chorionic gonadotropin (β-HCG)
* Biochemical abnormalities as indicated by liver function tests, and/or creatinine >1.5 times above upper limit of the normal range.
* Receiving any routine medications that may interfere with test drug metabolism that cannot be stopped one week prior to onset of study
* Evidence of urinary tract infection as indicated by an active urinary sediment (>6- 8 pus/neutrophil cells per field) or 3+ nitrate on dipstick. Individuals without a gross active sediment 1 or 2 plus nitrate or with 1 + protein will not be excluded. Similarly individuals with 1+ haemoglobin on dipstick or trace amount of blood in the will not be excluded.
* Lactose and/or gluten intolerance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-04-17 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06-04 (Actual)

PRIMARY OUTCOMES:
Drug Levels | up to 12 hours
  Five mil-liters of blood will be taken to test drug levels

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 (aggregate) | up to 1 year
  Following drug administration, a review of subjective symptoms will be performed.
Impact of treatment on Hematuria and Proteinuria | up to 7 days
  Urine samples will be collected to examine the the presence and amount of blood and protein in the urine.
Number worm nests | up to 1 year
  In those individuals with LF, an ultrasound examination will be performed to identify the number of adult worm nests both before treatment and after.
Impact of treatment on Liver Function + | up to 7 days
  Blood samples will be collected to examine the impact of treatment on the levels of ALT, AST in the subjects blood.
Impact of treatment on Hemoglobin Levels | up to 7 days
  Blood samples will be collected to examine the impact of treatment on the levels of Hemoglobin in the subjects blood.
Impact of treatment on White Blood Cells | up to 7 days
  Blood samples will be collected to examine the impact of treatment on the levels of white blood count in subjects blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Agboville District Hospital, Agbobille, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Andrade LD, Medeiros Z, Pires ML, Pimentel A, Rocha A, Figueredo-Silva J, Coutinho A, Dreyer G. Comparative efficacy of three different diethylcarbamazine regimens in lymphatic filariasis. Trans R Soc Trop Med Hyg. 1995 May-Jun;89(3):319-21. doi: 10.1016/0035-9203(95)90561-8. PMID 7660449
- [Background] Awadzi K, Edwards G, Duke BO, Opoku NO, Attah SK, Addy ET, Ardrey AE, Quartey BT. The co-administration of ivermectin and albendazole--safety, pharmacokinetics and efficacy against Onchocerca volvulus. Ann Trop Med Parasitol. 2003 Mar;97(2):165-78. doi: 10.1179/000349803235001697. PMID 12803872
- [Background] Awadzi K, Edwards G, Opoku NO, Ardrey AE, Favager S, Addy ET, Attah SK, Yamuah LK, Quartey BT. The safety, tolerability and pharmacokinetics of levamisole alone, levamisole plus ivermectin, and levamisole plus albendazole, and their efficacy against Onchocerca volvulus. Ann Trop Med Parasitol. 2004 Sep;98(6):595-614. doi: 10.1179/000349804225021370. PMID 15324466
- [Background] Bolla S, Boinpally RR, Poondru S, Devaraj R, Jasti BR. Pharmacokinetics of diethylcarbamazine after single oral dose at two different times of day in human subjects. J Clin Pharmacol. 2002 Mar;42(3):327-31. doi: 10.1177/00912700222011247. PMID 11865970
- [Background] Dominguez-Vazquez A, Taylor HR, Greene BM, Ruvalcaba-Macias AM, Rivas-Alcala AR, Murphy RP, Beltran-Hernandez F. Comparison of flubendazole and diethylcarbamazine in treatment of onchocerciasis. Lancet. 1983 Jan 22;1(8317):139-43. doi: 10.1016/s0140-6736(83)92753-8. PMID 6130195
- [Background] El Setouhy M, Ramzy RM, Ahmed ES, Kandil AM, Hussain O, Farid HA, Helmy H, Weil GJ. A randomized clinical trial comparing single- and multi-dose combination therapy with diethylcarbamazine and albendazole for treatment of bancroftian filariasis. Am J Trop Med Hyg. 2004 Feb;70(2):191-6. PMID 14993632
- [Background] Geary TG. Ivermectin 20 years on: maturation of a wonder drug. Trends Parasitol. 2005 Nov;21(11):530-2. doi: 10.1016/j.pt.2005.08.014. Epub 2005 Aug 26. PMID 16126457
- [Background] Hooper PJ, Chu BK, Mikhailov A, Ottesen EA, Bradley M. Assessing progress in reducing the at-risk population after 13 years of the global programme to eliminate lymphatic filariasis. PLoS Negl Trop Dis. 2014 Nov 20;8(11):e3333. doi: 10.1371/journal.pntd.0003333. eCollection 2014 Nov. PMID 25411843
- [Background] Horton J. Albendazole: a review of anthelmintic efficacy and safety in humans. Parasitology. 2000;121 Suppl:S113-32. doi: 10.1017/s0031182000007290. PMID 11386684
- [Background] Horton J. Albendazole: a broad spectrum anthelminthic for treatment of individuals and populations. Curr Opin Infect Dis. 2002 Dec;15(6):599-608. doi: 10.1097/00001432-200212000-00008. PMID 12821837
- [Background] Horton J. The development of albendazole for lymphatic filariasis. Ann Trop Med Parasitol. 2009 Oct;103 Suppl 1:S33-40. doi: 10.1179/000349809X12502035776595. PMID 19843396
- [Background] Horton J, Witt C, Ottesen EA, Lazdins JK, Addiss DG, Awadzi K, Beach MJ, Belizario VY, Dunyo SK, Espinel M, Gyapong JO, Hossain M, Ismail MM, Jayakody RL, Lammie PJ, Makunde W, Richard-Lenoble D, Selve B, Shenoy RK, Simonsen PE, Wamae CN, Weerasooriya MV. An analysis of the safety of the single dose, two drug regimens used in programmes to eliminate lymphatic filariasis. Parasitology. 2000;121 Suppl:S147-60. doi: 10.1017/s0031182000007423. PMID 11386686
- [Derived] Alshehri A, Chhonker YS, Bala V, Edi C, Bjerum CM, Koudou BG, John LN, Mitja O, Marks M, King CL, Murry DJ. Population pharmacokinetic model of ivermectin in mass drug administration against lymphatic filariasis. PLoS Negl Trop Dis. 2023 Jun 1;17(6):e0011319. doi: 10.1371/journal.pntd.0011319. eCollection 2023 Jun. PMID 37262040
- [Derived] Bala V, Chhonker YS, Alshehri A, Edi C, Bjerum CM, Koudou BG, King CL, Murry DJ. Population Pharmacokinetics of Diethylcarbamazine in Patients with Lymphatic Filariasis and Healthy Individuals. Antimicrob Agents Chemother. 2021 Sep 17;65(10):e0031721. doi: 10.1128/AAC.00317-21. Epub 2021 Jul 26. PMID 34310218
- [Derived] Edi C, Bjerum CM, Ouattara AF, Chhonker YS, Penali LK, Meite A, Koudou BG, Weil GJ, King CL, Murry DJ. Pharmacokinetics, safety, and efficacy of a single co-administered dose of diethylcarbamazine, albendazole and ivermectin in adults with and without Wuchereria bancrofti infection in Cote d'Ivoire. PLoS Negl Trop Dis. 2019 May 20;13(5):e0007325. doi: 10.1371/journal.pntd.0007325. eCollection 2019 May. PMID 31107869